CLINICAL TRIAL: NCT05461703
Title: "Efficacy of a School-based Obesity Prevention Program Delivery by Nutrition and Physical Activity Advanced Students or School Teachers on the BMI Z-score and Body Fat at 6 Months of Mexican Children: a Cluster Randomized Controlled Trial"
Brief Title: Efficacy of a School-based Obesity Prevention Program in Mexican Schoolchildren: Cluster Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Sonora (Other)
Collaborators: Centro de Investigación en Alimentación y Desarrollo A.C. (Other); Instituto Nacional de Geriatria, Mexico (Other Government); Universidad de León (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Full-time professor and researcher, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PNP02
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Obesity
Keywords: Obesity prevention; School-based program; Nutrition education; Physical activity; Cluster randomized controlled trial
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial. The study will be conducted in two phases. The first will be a 6-month pilot study with a follow-up at 8 months (after the summer holidays) and the second a definitive study of 6 months with a follow-up at 8 and 12 months. The study will consist of three parallel, three-arm groups with a 1:1:1 allocation ratio.
Who Masked: Investigator
Masking Description: The person in charge of the allocation of the schools will be blinded. The outcome assessors will also be blinded to the group allocation of the schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Planet Nutrition Program (PNP) implemented by nutrition and physical activity advanced students (Experimental): The PNP consists of:
  Nutrition education sessions: Nutrition advanced students of the University of Sonora will provide 1 face-to-face group class of one hour per week. The PNP handbook will be used to bring the different topics and dynamics to reinforce learning. The program will be focused on establishing some health-related goals.
  Physical activity sessions: Three classes of 1 hour per week will be implemented by physical activity advanced students of the University of Sonora, independent of the school's curricular physical activity classes. A physical activity handbook designed by the study team will be used. Children will work on developing different skills.
  Parents participation: They will receive one printed brochure with nutrition topics weekly. Also, they will be asked for their Facebook user (to create a private group) or the email to upload the information of the brochure and other didactic materials. Nutrition students will be in charge of providing the information.
  Interventions: Behavioral: Planet Nutrition Program
- Planet Nutrition (PNP) implemented by school teachers (Experimental): The PNP consists of:
  Nutrition education sessions: Fourth grade school teachers will provide 1 face-to-face group class of one hour per week. The PNP handbook will be used to bring the different topics and dynamics to reinforce learning. The program will be focused on establishing some health-related goals.
  Physical activity sessions: Three classes of 1 hour per week will be implemented by physical activity advanced students of the University of Sonora, independent of the school's curricular physical activity classes. A physical activity handbook designed by the study team will be used. Children will work on developing different skills.
  Parents participation: They will receive one printed brochure with nutrition topics weekly. Also, they will be asked for their Facebook user (to create a private group) or the email and upload the information of the brochure and other didactic materials. School teachers will be in charge of providing the information.
  Interventions: Behavioral: Planet Nutrition Program
- Control Group (No Intervention): Scholars of this group will continue with their normal school nutrition and physical activity classes. At the end of the study they will have access to the program materials through a web page.

INTERVENTIONS:
Behavioral: Planet Nutrition Program — It is a 6-month school-based obesity prevention program that includes: nutrition education sessions, physical activity and family participation.
  Arms: Planet Nutrition (PNP) implemented by school teachers; Planet Nutrition Program (PNP) implemented by nutrition and physical activity advanced students

SUMMARY:
There is evidence that obesity prevention programs show positive effects on obesity and lifestyle parameters. However, the effect of the programs delivered by different implementers is unknown, and in Mexico, the available studies present methodological limitations. The aim of this study is to evaluate the feasibility and efficacy of a school-based obesity prevention program implemented by nutrition and physical activity advanced students compared to a control group and implemented by school teachers compared to a control group of Mexican schoolchildren. This is a cluster randomized controlled trial. Schoolchildren from different public schools in Hermosillo , Sonora will be invited to participate. The schools will be randomly assigned to one option:1) the Planet Nutrition Program (PPN) delivered by advanced students, 2) PPN by school teachers, or 3) a control group. A 6-month pilot study with a follow-up at 8 months (after the summer holidays), followed by a definitive study with a follow-up at 8 and 12 months will be conducted.The intervention will consist of nutrition education sessions, physical activity, and the provision of nutrition information for parents. The BMI Z-score, body fat, other obesity, and lifestyle parameters will be evaluated at baseline and at the end of the study. A mixed effects model will be used to evaluate the differences between the groups. The investigators expect that the program could be a model of obesity prevention with a high potential for dissemination in Mexican schools.

DETAILED DESCRIPTION:
This is a cluster randomized controlled trial. The study will be conducted in two phases. The first phase will be a 6-month pilot study with a follow-up at 8 months (after the summer holidays) to evaluate the feasibility: of retention, adherence, acceptability, and fidelity (Eldridge et al, 2010). The second will be a definitive study of 6 months with a follow-up at 8 and 12 months to evaluate the efficacy. The study will consist of three parallel, three-arm groups with a 1:1:1 allocation ratio.

To perform the protocol of the study, the SPIRIT 2013 guide was followed. The study was approved by the Research Ethics Committee of the University of Sonora Department of Nursing (EPD-007-2022).

Fifteen public schools (300 to 450 students) from Hermosillo, Sonora, Mexico will be conveniently invited to participate in the pilot study. The sample size was determined based on the capacity of providing the program and on finding possible positive effects on the variables of interest . The calculation of the sample size is not essential in a pilot study, where its main objective is to know the feasibility of the intervention and information regarding the response variables to later carry out the sample size calculation for a future definitive trial (Eldridge, 2016).

Once the informed consent and assent have been signed by the parents and children (respectively), the baseline measurements will be made over 4 weeks. The schools and participants that meet the inclusion/exclusion criteria will be randomly assigned to one of the three arms. 1). Planet Nutrition Program (PNP) implemented by nutrition and physical activity advanced students (studying the last semesters of the degree or who have completed subjects but do not have the degree), 2). PNP implemented by school teachers and 3). a control group. An independent person from the recruitment and the intervention will perform the random allocation of the schools. This will be stratified by socioeconomic level. The random number sequence will be generated using the software "Research Randomizer" https://randomizer.org/.

The baseline characteristics will be analyzed among groups, and an ANOVA analysis will be used for the quantitative variables, and a chi-square test for the categorical outcomes in order to assure that groups are similar in all variables. If there are significant differences among groups at baseline, an adjustment will be made in the analysis. To evaluate the differences between groups in the change of the BMI Z-score, body fat, and the other secondary variables at the beginning and at the end of the intervention, a mixed model will be used to consider the effect between groups and within groups. All analyzes will be performed by the intention to treat. If data is not obtained for any reason or subjects were excluded due to a protocol violation, they will be replaced by their baseline measurement. The R studio software will be used to perform the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Schools:

  * school directors and teachers wish to participate.
  * availability of space for physical activity classes.
  * the school has at least 20 children per 4th-grade group.
* Schoolchildren:

  -be a 4th grade student (9 to 11 years old).
* Implemeters:

  * receive 80% of the program training.
  * respond satisfactorily to a questionnaire that tests knowledge of the program

Exclusion Criteria:

* Schools: participating in another similar study.
* Schoolchildren: Having a personal condition that prevents physical activity or a condition that parents consider should not involve the child.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Retention assessed by the number of participants/schools that complete the study (more information in the description). | At 6 months
  This variable will be obtained with the number of schools and participants that complete the final measurements of the study. At 6 months, retention of participants and schools >80% will be considered excellent, >50-80 moderate, and <50 low retention.
Adherence evaluated with the number of sessions attended by the participants (more information in the description). | At 6 months.
  It will be evaluated with the number of attended sessions by schoolchildren and parents of the intervention groups. At 6 months, the attendance at program activities >80 will be considered excellent, >50-80 moderate, and <50 low attendance.
Fidelity evaluated with the number of sessions provided by the implementers (more information in the description). | At 6 months.
  This will be evaluated with a questionnaire to ask implementers about the number of sessions and workshops implemented. Excellent fidelity to the study activities will be considered when ≥ 60% of the program is delivered, <60-40% moderate, and <40 % low.
Acceptability of the intervention assessed by a questionnaire of the research team (information in the description). | At 6 months.
  The variable will be obtained with a questionnaire designed by the research group (not validated), applied to the children and parents of the intervention groups to qualify the program and materials. Also, to know about the benefits obtained with the program. A questionnaire will be provided to implementers to indicate their acceptance of the program and barriers to provide the sessions. It will be considered as good acceptance with a score of > 8-10 points, moderate acceptance > 5-8 points, and low acceptance ≤5 points.
Change in the BMI Z-score | Baseline, at 6 months, 8 months (after summer holidays), and for the definitive trial: baseline, 6 months, 8 months and after the 12 months of follow-up.
  It will be the primary outcome for the definitive study. The BMI Z-score will be obtaining with the weight, height, gender and date of birth of the children, using the "Anthro Plus" software, which utilize the WHO reference tables (WHO,2007). The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Change in Body fat | Baseline, at 6 months, 8 months (after summer holidays), and for the definitive trial: baseline, 6 months, 8 months and after the 12 months of follow-up.
  It will be the primary outcome for the definitive study. The tetrapolalar electrical bioimpedance method will be used to obtain the resistance and reactance values. The measurement will be carried out with a bioimpedance electrical equipment, RJL Quantum II, following the methodology used by Ramírez et al. With the data obtained, an equation designed to estimate fat-free mass in Mexican children will be used (Ramírez et al,2012). The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.

SECONDARY OUTCOMES:
Change in Weight | Baseline, at 6 months and 8 months (after summer holidays), and for the definitive trial: baseline, 6 months, and after the 8 months and 12 months of follow-up.
  A TANITA SC-240 scale will be used to measure the body weight. The measurement will be take without shoes and accessories with light clothes. Children will stand in the center of the scale with their feet separated and arms at their sides. Measurement will be used to obtain the BMI Z-score (Gibson, 1990). The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Change in Waist circumference | Baseline and 6 months.
  A metallic anthropometric tape (Lufkin Executive Thineline W606PMM) will be used, taking the umbilical scar as measurement reference and in a standing position (Gibson,1990). The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Change in Relative fat mass | Baseline and 6 months.
  This is an estimator of total body fat. The relative fat mass will be estimated using a formula validated with American children aged 8 to 14 years. Data of waist circumference (cm), height (cm) and sex will be used (Woolcott et al,2019). The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Change in Food consumption | Baseline and 6 months.
  Some questions from the semi-quantitative food frequency questionnaire (FFQ) from the National Health and Nutrition Survey will be used.(Shamah-levy et al,2016).We will asked about the frequency of consumption of ultra-processed foods (sweet beverages, fried foods, cakes and cookies) and healthy foods (fruits, vegetables and water) in the previous 7 days. For each food, the size of the portion consumed will be asked, considering an average portion established in the FFQ. The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Change in Physical activity and sedentary behavior | Baseline and 6 months.
  The questions on physical activity and sedentary lifestyle will be used from the questionnaire, "The Health Behavior in School-Age Children" (HBSC) (Currie et al,2014). It includes the days and the time dedicated to physical activity and sedentary activities during the last 7 days in sedentary activities during the week and at the weekend. The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Chane in Quality of life, assessed by PedsQL (more information in the description) | Baseline and 6 months.
  The PedsQL™ questionnaire (Pediatric Quality of Life Inventory) will be used. This generic health status instrument assesses the frequency of problems experienced in the past month in physical, emotional, social, and school functioning. Responses are on a 5-point likert scale (never = 0 to always = 4). The score for each item is inverted and converted to a linear scale from 0 to 100, a higher score indicates a better quality of life (Varni et al,2001).The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.
Nutrition knowledge | Baseline and 6 months.
  A questionnaire designed by the study team will be used to assess knowledge on nutrition issues. It consists of 32 questions about nutrition and health. They will be evaluated on a scale from 0 to 10, the more correct answers, the higher the score.The change in the outcome will be obtained by subtracting the value obtained at the final measurement from the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz Zavala, PhD, Principal Investigator — Universidad de Sonora
Locations (1):
- Public Schools, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization (WHO). Obesity and Overweight. [Internet]. 2018 [cited 2019 Oct 10]. Available from: https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Shamah-Levy T, Vielma-Orozco E, Heredia-Hernández O, Romero-Martínez M, Mojica-Cuevas J C-NL, Santaella-Castell JA R-DJ. Encuesta Nacional de Salud y Nutrición 2018-19: Resultados Nacionales. [Internet]. Cuernavaca, México; 2020. Available from: https://ensanut.insp.mx/encuestas/ensanut2018/informes.php
- [Background] Obesity Evidence Hub. Obesity trends in children globally [Internet]. 2021 [cited 2021 Nov 20]. Available from: https://www.obesityevidencehub.org.au/collections/trends/children-global-context
- [Background] Sharma V, Coleman S, Nixon J, Sharples L, Hamilton-Shield J, Rutter H, Bryant M. A systematic review and meta-analysis estimating the population prevalence of comorbidities in children and adolescents aged 5 to 18 years. Obes Rev. 2019 Oct;20(10):1341-1349. doi: 10.1111/obr.12904. Epub 2019 Jul 24. PMID 31342672
- [Background] Lambrinou CP, Androutsos O, Karaglani E, Cardon G, Huys N, Wikstrom K, Kivela J, Ko W, Karuranga E, Tsochev K, Iotova V, Dimova R, De Miguel-Etayo P, M Gonzalez-Gil E, Tamas H, Jancso Z, Liatis S, Makrilakis K, Manios Y; Feel4Diabetes-study group. Effective strategies for childhood obesity prevention via school based, family involved interventions: a critical review for the development of the Feel4Diabetes-study school based component. BMC Endocr Disord. 2020 May 6;20(Suppl 2):52. doi: 10.1186/s12902-020-0526-5. PMID 32370795
- [Background] WHO. Population-based approaches to childhood obesity prevention [Internet]. Geneva, Switzerland; 2012. Available from: https://www.who.int/dietphysicalactivity/childhood/WHO_new_childhoodobesity_PREVENTION_27nov_HR_PRINT_OK.pdf
- [Background] Pulimeno M, Piscitelli P, Colazzo S, Colao A, Miani A. School as ideal setting to promote health and wellbeing among young people. Health Promot Perspect. 2020 Nov 7;10(4):316-324. doi: 10.34172/hpp.2020.50. eCollection 2020. PMID 33312927
- [Background] Brown T, Moore TH, Hooper L, Gao Y, Zayegh A, Ijaz S, Elwenspoek M, Foxen SC, Magee L, O'Malley C, Waters E, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2019 Jul 23;7(7):CD001871. doi: 10.1002/14651858.CD001871.pub4. PMID 31332776
- [Background] Singhal J, Herd C, Adab P, Pallan M. Effectiveness of school-based interventions to prevent obesity among children aged 4 to 12 years old in middle-income countries: A systematic review and meta-analysis. Obes Rev. 2021 Jan;22(1):e13105. doi: 10.1111/obr.13105. Epub 2020 Jul 28. PMID 32725780
- [Background] Aceves-Martins M, Lopez-Cruz L, Garcia-Botello M, Gutierrez-Gomez YY, Moreno-Garcia CF. Interventions to Prevent Obesity in Mexican Children and Adolescents: Systematic Review. Prev Sci. 2022 May;23(4):563-586. doi: 10.1007/s11121-021-01316-6. Epub 2021 Nov 2. PMID 34725762
- [Background] Ramirez-Rivera DL, Martinez-Contreras T, Villegas-Valle RC, Henry-Mejia G, Quizan-Plata T, Haby MM, Diaz-Zavala RG. Preliminary Results of the Planet Nutrition Program on Obesity Parameters in Mexican Schoolchildren: Pilot Single-School Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jan 18;18(2):790. doi: 10.3390/ijerph18020790. PMID 33477722
- [Background] Ramírez-Rivera DL, Martínez-Contreras T, Henry-Mejia G, Ruelas AL, Quizán-Plata T, Esparza-Romero J, Díaz-Zavala RG. Efecto de una intervención en línea de cambio en el estilo de vida sobre el puntaje zIMC de escolares mexicanos: protocolo de ensayo controlado aleatorizado piloto cegado a evaluadores durante la pandemia por COVID-19. Rev Esp Nutr Hum Diet 2021;25.
- [Background] Diaz-Zavala RG, Castro-Cantu MF, Valencia ME, Alvarez-Hernandez G, Haby MM, Esparza-Romero J. Effect of the Holiday Season on Weight Gain: A Narrative Review. J Obes. 2017;2017:2085136. doi: 10.1155/2017/2085136. Epub 2017 Jul 4. PMID 28744374
- [Background] Franckle R, Adler R, Davison K. Accelerated weight gain among children during summer versus school year and related racial/ethnic disparities: a systematic review. Prev Chronic Dis. 2014 Jun 12;11:E101. doi: 10.5888/pcd11.130355. PMID 24921899
- [Background] Fernandez ME, Ruiter RAC, Markham CM, Kok G. Intervention Mapping: Theory- and Evidence-Based Health Promotion Program Planning: Perspective and Examples. Front Public Health. 2019 Aug 14;7:209. doi: 10.3389/fpubh.2019.00209. eCollection 2019. PMID 31475126
- [Background] Murimi MW, Moyeda-Carabaza AF, Nguyen B, Saha S, Amin R, Njike V. Factors that contribute to effective nutrition education interventions in children: a systematic review. Nutr Rev. 2018 Aug 1;76(8):553-580. doi: 10.1093/nutrit/nuy020. PMID 29800311
- [Background] Universidad de Guadalaja. Pedirá AMFEN regular apertura de escuelas de Nutrición en México [Internet]. 2021. Available from: http://www.cualtos.udg.mx/noticia/pedira-amfen-regular-apertura-de-escuelas-de-nutricion-en-mexico.
- [Background] El País. Universidades que imparten Deportes [Internet]. 2021. Available from: https://elpais.com/especiales/2015/carreras-mexico/carrera/universidad/deportes.html
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] WHO. Growth Reference 5-19 years. BMI-for-age (5-19 years). [Internet]. 2007. Available from: https://www.who.int/growthref/en/
- [Background] Ramirez E, Valencia ME, Bourges H, Espinosa T, Moya-Camarena SY, Salazar G, Aleman-Mateo H. Body composition prediction equations based on deuterium oxide dilution method in Mexican children: a national study. Eur J Clin Nutr. 2012 Oct;66(10):1099-103. doi: 10.1038/ejcn.2012.89. Epub 2012 Jul 18. PMID 22805494
- [Background] Gibson R. Principles of Nutritional Assessment. New York: Oxford University Press; 1990.
- [Background] Woolcott OO, Bergman RN. Relative Fat Mass as an estimator of whole-body fat percentage among children and adolescents: A cross-sectional study using NHANES. Sci Rep. 2019 Oct 24;9(1):15279. doi: 10.1038/s41598-019-51701-z. PMID 31649287
- [Background] Shamah-Levy T, Cuevas-Nasu L, Rivera-Dommarco J, Hernández-Ávila M. Encuesta Nacional de Salud y Nutrición de Medio Camino 2016. (ENSANUT MC 2016) [Internet]. 2016. Available from: gob.mx/salud/documentos/encuesta-nacional-de-salud-y-nutricion-de-medio-camino-2016.
- [Background] Currie C, Inchley J, Molcho M, Lenzi M, Veselska Z, Wild F. Health Behaviour in School-aged Children (HBSC) study protocol: background , methodology and mandatory items for the 2013/14 survey [Internet]. 2014. Available from: http://www.hbsc.org
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499